CLINICAL TRIAL: NCT06996405
Title: EFFECT Diet - Cluster RCT and Qualitative Inquiry
Brief Title: Effect of Access to Dietary Intervention in a Dialysis Unit
Acronym: EFFECTdiet
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Steno Diabetes Center Sjaelland (Other Government); The Danish Kidney Association (Other); VIA University College (Other); The Danish Dietetic Association (Other)
Responsible Party: Principal Investigator, Anne Sofie Wendelboe Jørgensen, ph.d. student/ dietitian, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EFFECT diet
Record Dates: First submitted 2025-04-11; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Dialysis; Diabetes; Nutritional Status; Diet Therapy
Keywords: Dietary intervention; Dietitian
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutritional therapy (Active Comparator): Access to diet intervention
  Interventions: Other: Access to dietary treatment
- Usual care (No Intervention): Usual care. Referral to dietitian if needed

INTERVENTIONS:
Other: Access to dietary treatment — Dietary treatment using current nutrition guidelines, dialogic communication and Nutrition Care Process repeatedly by weekly access to a dietitian for four month.
  Arms: Nutritional therapy

SUMMARY:
Objective:

The aim of this study is to explore the effect of access to individual dietary counselling by a dietitian in the dialysis unit on biochemical values (phosphorus and potassium), diet, nutritional status, quality of life (QoL) and health literacy (HL).

Hypothesis: Having access to a dietitian can better laboratory values and affect dietary intake, nutritional status, QoL and HL in a positive matter.

Method:

Pilot cluster RCT study in three the dialysis units in Region Zealand. Clustering of people on dialysis the same day to either intervention or control group. The groups is expected to be similar regarding clinical characteristics.

Primary outcome: Change in average p-phosphate Secondary outcomes: Change in average p-potassium, number of phosphate binders, number of potassium binders, HeartDiet-score, Nutritional Status, Adherence to diet (End Stage Renal Disease Adherence Questionnaire), Quality of life (Kidney Disease Quality of Life Short Form) and Health literacy (Health Literacy Questionnaire)

Intervention:

The intervention group receives an initial individual dietary interview, monthly follow-up and weekly access to a dietitian in the dialysis unit for four months. The control group receives usual care with referral to a dietitian when needed.

DETAILED DESCRIPTION:
Objective:

The aim of this study is to explore the effect of access to individual dietary counselling by a dietitian in the dialysis unit on biochemical values (phosphorus and potassium), diet, nutritional status, quality of life (QoL) and health literacy (HL).

Research question:

What is the effect of access to dietary treatment in people receiving dialysis treatment on biochemical values (phosphorus and potassium), diet, nutritional status, quality of life and health literacy? Hypothesis: Having access to a dietitian can better laboratory values and affect dietary intake, nutritional status, QoL and HL in a positive matter.

Method:

Pilot cluster RCT study in the dialysis units in Holbæk and Slagelse in Region Zealand, Denmark. Clustering of people on dialysis the same day to either intervention or control group. The groups is expected to be similar regarding clinical characteristics. A pilot project will be conducted in 2024 in the dialysis units in Slagelse and Holbæk.

Data collection:

Both groups:

* Patient characteristics (at the beginning of project): Age and gender, height, medical diagnosis, socioeconomic data (income, job, education, partner status) and dialysis vintage.
* Clinical Data (before and after the intervention, and at 6 and 12 month after the intervention period): Biochemical values (phosphate, potassium, urea, albumin, PTH), anthropometric measures (dry weight, actual weight), medication, ultrafiltration, and number of contacts with dietitian.
* Questionnaires and tests (collected before and after the intervention): Body composition (fat, fat-free mass, water), Nutritional status, Intake (HeartDiet Questionnaire), Quality of Life (KDQOL-SF), Health Literacy (HLQ), and previous dietary treatment.

Primary outcome: Change in average p-phosphate Secondary outcomes: Change in average p-potassium, number of phosphate binders, number of potassium binders, HeartDiet-score, Nutritional Status (nutritional screening), Adherence to diet (End Stage Renal Disease Adherence Questionnaire, ESRD-AQ-score), Quality of life (Kidney Disease Quality of Life Short Form, KDQOL-SF-score) and Health literacy (Health Literacy Questionnaire, HLQ-score)

Intervention:

The intervention group receives an initial individual dietary interview, monthly follow-up and weekly access to a dietitian in the dialysis unit for four months.

The individualized dietary treatment based on the patient's preferences and needs according to the Nutrition Care Process. It is carried out according to the practical guidelines from the Danish Dietetic Association on dietary treatment of chronic kidney disease. The dietary treatment uses a dialogic and person-centered approach The intervention is described in the protocol using the TIDieR framework. The control group receives usual care with referral to a dietitian when needed.

Statistics:

The average phosphorus level and standard deviation after a diet intervention was 1.58 ± 0.32 mmol/l, therefore using 0.32 mmol/l in calculation of sample size. An implementation of guidelines and a systematic review showed a difference in phosphosus levels between intervention and control group of 0.23 and 0.30 mmol/l respectively.

Calculation of sample size using "Sample Size Calculator (clincalc.com)". Using the values mentioned above, a power of 80% and a significance of 5% shows a sample size of 18-30 people in each group to show a significant change in phosphorus levels.

Comparison of changes in average values using unpaired t-test, including endpoints of p-phosphorous and p-potassium, QoL-score and health literacy score. For dichotomous endpoints such as nutritional score, comparison of the percentage of the groups within and without specific limits. Data analysis with intention-to-treat and statistical calculations by a person not familiar with the groups.

ELIGIBILITY:
Inclusion criteria:

* Able to understand Danish
* Chronic dialysis treatment (min. 3 month)

Exclusion criteria:

* Dementia
* Not able to sign a consent form
* Expected short duration of life, eg. terminal cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Average phosphate | At baseline and after 5 month at the end of the intervention period (last phosphate value before termination of intervention), and 6 and 12 month post-intervention (counting from last day of intervention)
  Difference in average phosphate-level between groups

SECONDARY OUTCOMES:
Phosphate-level | At baseline and after 5 month at the end of the intervention period (last phosphate value before termination of intervention), and 6 and 12 month post-intervention (counting from last day of intervention)
  Number of patients with phosphate-level within range
Phosphate-level | At baseline and after 5 month at the end of the intervention period (last phosphate value before termination of intervention), and 6 and 12 month post-intervention (counting from last day of intervention)
  Number of patients experiencing a increase or decrease in phosphate to/ from range
Phosphate binders | At baseline, changes within the intervention period, after 5 month at the end of the intervention period, and 6 and 12 month after the last day of the intervention
  Change in numbers of prescribed phosphate binders
Average potassium | At baseline and after 5 month at the end of the intervention period (last potassium value before termination of intervention), and 6 and 12 month post-intervention (counting from last day of intervention)
  Difference in average potassium-level between groups
Potassium-level | At baseline and after 5 month at the end of the intervention period (last potassium value before termination of intervention), and 6 and 12 month post-intervention (counting from last day of intervention)
  Number of patients with potassium-level within range
Potassium-level | At baseline and after 5 month at the end of the intervention period (last potassium value before termination of intervention), and 6 and 12 month post-intervention (counting from last day of intervention)
  Number of patients experiencing a increase or decrease in potassium to/ from range
Potassium binders | At baseline, changes within the intervention period, after 5 month at the end of the intervention period, and 6 and 12 month after the last day of the intervention
  Change in numbers of prescribed potassium binders
Nutritional Status | At baseline and after 5 month at the end of the intervention period
  Nutritional screening according to Nutritional Risk Screening (NRS-2002)
Nutritional intake | At baseline and after 5 month at the end of the intervention period
  Nutritional intake collected using the food frequency questionnaire HeartDiet
Quality of Life-score | At baseline and after 5 month at the end of the intervention period
  Quality of Life-score using the questionnaire Kidney Disease Quality of Life Short Form (KDQOL-SF)
Adherence-score | At baseline and after 5 month at the end of the intervention period
  Adherence-score using the questionnaire End Stage Renal Disease Adherence Questionnaire (ESRD-AQ)
Symptom-score | At baseline and after 5 month at the end of the intervention period
  Symptom-score using the questionnaire The Integrated Palliative Outcome Scale - Renal (IPOS-RENAL)
Health Literacy Questionnaire-score | At baseline and after 5 month at the end of the intervention period
  Health Literacy Questionnaire-score using the questionnaire Health Literacy Questionnaire (HLQ)

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Wendelboe, Principal Investigator — Zealand University Hospital
Locations (3):
- Denmark (3):
  - Holbæk Dialysis Unit, Holbæk
  - Næstved Dialysis Unit, Næstved
  - Slagelse Dialysis Unit, Slagelse

IPD SHARING:
Plan to Share IPD: No